CLINICAL TRIAL: NCT04956302
Title: A Phase I Study of Panobinostat in Combination With Daratumumab, Bortezomib, and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Panobinostat in Combination With Daratumumab, Bortezomib and Dexamethasone for the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Abdullah Khan (Other)
Responsible Party: Sponsor-Investigator, Abdullah Khan, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21005; NCI-2021-04261 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (panobinostat, daratumumab, bortezomib, dexa) (Experimental): Patients receive panobinostat PO QD on days 1, 3, 5, 15, 17, 19, daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles, bortezomib SC on days 1, 8, 15, 22 and dexamethasone PO (IV on days of daratumumab and hyaluronidase-fihj administration) QD on days 1, 8, 15, 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Panobinostat Lactate

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Daratumumab and Hyaluronidase-fihj — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Panobinostat Lactate — Given PO
  Other Names: Farydak

SUMMARY:
This phase I trial studies the possible benefits and side effects of adding panobinostat to a combination of daratumumab, bortezomib and dexamethasone in treating patients with multiple myeloma that has come back (relapsed) or has not responded to treatment (refractory). Panobinostat may stop or slow multiple myeloma by blocking the growth of new blood vessels necessary for cancer growth. Giving panobinostat in combination with daratumumab, bortezomib and dexamethasone may work better in treating relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of Farydak (panobinostat lactate)/Darzalex Faspro (daratumumab and hyaluronidase-fihj)/Velcade (bortezomib)/dexamethasone (FDVd) in patients with relapsed/refractory multiple myeloma (RRMM) who have previously received one line of therapy including lenalidomide or cyclophosphamide, bortezomib (V) or other proteasome inhibitor (PI), with or without autologous stem cell transplant (ASCT).

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) (per International Myeloma Working Group [IMWG] criteria) of FDVd.

II. Determine the time to response (TTR). III. Determine the duration of response (DOR). IV. Determine the progression-free survival (PFS) at 1 year. V. Determine the overall survival (OS) at 1 year.

CORRELATIVE OBJECTIVES:

I. Baseline and end of-study plasma cell expression of CD38. II. Changes in lymphocyte subsets with therapy. III. Baseline and end-of study analysis of total number and ratio of regulatory T cells (Tregs) with CD38+ expression.

IV. Check minimal residual disease (MRD) negativity rates by next generation sequencing in patients who attain and maintain very good partial response (VGPR) or better for at least three months.

OUTLINE: This is a dose-escalation study of panobinostat.

Patients receive panobinostat orally (PO) once daily (QD) on days 1, 3, 5, 15, 17, 19, daratumumab and hyaluronidase-fihj subcutaneously (SC) on days 1, 8, 15, 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles, bortezomib SC on days 1, 8, 15, 22 and dexamethasone PO (intravenously [IV] on days of daratumumab and hyaluronidase-fihj administration) QD on days 1, 8, 15, 22. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up on days 30 and 60.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 years of age with evidence of relapsed or refractory disease as defined by IMWG criteria and measurable disease as defined by any of the following:

  * Serum M-protein >= 0.5 g/dl (>= 10 g/l)
  * Urine monoclonal protein >= 200 mg/24h
  * Involved free light chain (FLC) level >= 10mg/dl (>= 100mg/l) and an abnormal serum free light chain ratio (< 0.26, or > 1.65)
* Patients must have had at least 1 prior line of therapy including lenalidomide or cyclophosphamide, V or other PI, with or without ASCT

  * Patients with progressive disease (PD) as best response on V are excluded
  * Patients with PD on D-based therapy may be eligible at the discretion of the treating physician
* Refractory (progressed on or within 120 days of treatment) to their last treatment

  * Patients must be off last treatment for at least 2 weeks by the beginning of treatment on this protocol
* Hemoglobin >= 7g/dL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 70,000/uL

  * If plasma cell percentage on bone marrow biopsy aspirate or core is > 30%, platelet requirement will be adjusted to 50,000/ul
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/alkaline phosphatase < 2 x the upper limit of normal (ULN)
* Serum creatinine < 2mg/dL or calculated creatinine clearance of >= 30ml/min using Modification of Diet in Renal Disease Study (MDRD) formula
* Left ventricular ejection fraction >= 30%; baseline echocardiogram (ECHO) is not required
* No uncontrolled arrhythmias
* No New York Heart Association class III-IV heart failure
* 12-lead electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of =< 450 msec
* Patient must be able to swallow capsule or tablet
* Patients must provide informed consent
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of < 2
* Women of child bearing potential (WOCBP) must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing and continue to 6 months after study treatment ending. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy
* Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy
* A negative pregnancy test will be required for all WOCBP within 24 hours before starting treatment drugs
* Breast feeding is not permitted
* Male patients must agree to use an adequate method of contraception (latex or synthetic condom) for the duration of the study and up to 6 months after study treatment ending

  * Criteria also applies to azoospermic males
* Males should refrain from sperm donation during this time and continue for 6 months after study treatment ending

Exclusion Criteria:

* Patients with active (untreated or relapsed) central nervous system (CNS) metastasis of myeloma
* Patients with Waldenstrom macroglobulinemia, primary amyloid light-chain (AL) amyloidosis, primary plasma cell leukemia, or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome

  * Patients with secondary plasma cell leukemia are permitted
* Patients with peripheral neuropathy > National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Patients receiving concurrent corticosteroids at the time protocol therapy is initiated other than for physiologic maintenance treatment
* Concurrent use of complementary or alternative medicines that would confound the interpretation of toxicities and antitumor activity of the study drugs
* Patients with known allergies, hypersensitivity, or intolerance to panobinostat, daratumumab, or bortezomib
* Unacceptable respiratory risk factors defined by any one of the following criteria:

  * Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) less than 50% of predicted normal
  * Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Unacceptable cardiac risk factors defined by any of the following criteria:

  * Patients with congenital long QT syndrome
  * Any history of ventricular fibrillation or torsade de pointes
  * Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm)
  * Left ventricular ejection fraction < 30%
* Patients who have received targeted or investigational agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is shorter) and who have not recovered from side effects of those therapies
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with active hepatitis B (defined as hepatitis B virus surface antigen positive [HBsAg+]); HBV screening is required prior to beginning therapy

  * Patients with prior hepatitis B vaccine are permitted (defined as hepatitis B virus surface antigen negative [HBsAg-], hepatitis B virus surface antibody positive [Anti-HBs+], hepatitis B virus core antibody negative (Anti-HBc-])
  * Non-active hepatitis B (HBsAg-, Anti-HBs+, hepatitis B virus core antibody positive [Anti-HBc+]) may only be enrolled following approval by the sponsor after consideration of risk of reactivation (additional screening and monitoring for hepatitis B and consultation with a liver disease specialist may be required)
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled

  * Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from a prior malignancy for >= 3 yrs, and are considered by their physician to be less than 30% risk of relapse
* Patients with a history of gastrointestinal surgery or other procedure that might, in the opinion of the investigator(s), interfere with the absorption or swallowing of the study drugs
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff
* Any other medical condition, including mental illness or substance abuse, deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose | End of cycle 1 (1 cycle = 28 days)
  A standard "3+3" design will be used to determine the safe and tolerable dose level.
Incidence of adverse events | Up to 3 years
  Assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

SECONDARY OUTCOMES:
Time to progression | From start of treatment until objective tumor progression, assessed up to 3 years
  Cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks.
Progression-free survival | From start of treatment until disease progression or death, assessed at 1 year
  Will be calculated using the Kaplan-Meier method. Will be calculated together with 95% confidence intervals, and log-rank test will be used for the comparison between patient subgroups.
Objective response rate (ORR) | Up to 3 years
  ORR will be defined as the total number of subjects whose best response is partial response (PR) or better divided by the number of patients. ORR will be reported overall as well as by dose level, with 95% binomial exact confidence intervals. Comparison of ORR among patient subgroups will be conducted using Fisher exact test.
Time to response | From start of treatment until measurement criteria are first met for PR, very good partial response, or complete response, assessed up to 3 years
  Cumulative incidence rates will be calculated and compared using Gray's test accounting for competing risks.
Duration of overall response | From the time measurement criteria are first met for partial response or better (whichever status is recorded first) until the first date of progressive disease or death, assessed up to 3 years
  Will be calculated using the Kaplan-Meier method. Will be calculated together with 95% confidence intervals, and log-rank test will be used for the comparison between patient subgroups.
Overall survival | From start of treatment to the date of his or her death, assessed at 1 year
  Will be calculated using the Kaplan-Meier method. Will be calculated together with 95% confidence intervals, and log-rank test will be used for the comparison between patient subgroups.

OTHER OUTCOMES:
Plasma cell expression of CD38 | Baseline up to 60 days
  Will be explored graphically (e.g. side-by-side boxplots) and with quantitative summaries, compared using Mann-Whitney test or Fisher exact test depending on the data type of expression data.
Changes in lymphocyte subsets with therapy | Baseline up to 60 days
Total number and ratio of regulatory T cells with CD38+ expression | Baseline up to 60 days
Minimal residual disease negativity rates by next generation sequencing in patients who attain and maintain very good partial response or better for at least three months | Baseline up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Khan, MBBS, MSc, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT04956302/ICF_000.pdf